CLINICAL TRIAL: NCT00627146
Title: Extension of Phase II Therapeutic Trial With a Humanized Non-Mitogenic CD3 (ChAgly CD3) Monoclonal Antibody in Recently Diagnosed Type 1 Diabetic Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AZ-VUB (Other)
Collaborators: KU Leuven (Other); Universiteit Antwerpen (Other); Erasme University Hospital (Other)
Responsible Party: Bart Keymeulen, Universitair Ziekenhuis Brussel
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BK-AntiCD3-02
Record Dates: First submitted 2008-02-22; First posted 2008-02-29 (Estimated); Last update posted 2008-09-29 (Estimated); Status verified 2008-09

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Diabetes Mellitus, type 1; ChAgly CD3
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — otelixizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- B (Placebo Comparator)
  Interventions: Drug: Placebo
- A (Active Comparator): ChAgly CD3
  Interventions: Drug: ChAgly CD3

INTERVENTIONS:
Drug: ChAgly CD3 — 6 days treatment 8mg/d intravenous
  Arms: A
Drug: Placebo — 6 days
  Arms: B

SUMMARY:
Compared to placebo, treatment with ChAgly CD3 has a beneficial effect on preservation of beta cell function and metabolic outcome in type 1 diabetic patients with recent clinical onset of disease that persists until 48 months after administration.

The investigators also hypothesize that in type 1 diabetic patients with recent clinical onset of disease compared to placebo, ChAgly CD3 will be safe and well tolerated between 18 and 48 months after administration, based on assessment of clinical and laboratory adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with Type 1 diabetes mellitus included in the phase II therapeutic trial with a humanized non-mitogenic CD3 monoclonal antibody (ChAgly CD3) at time of clinical diagnosis and who agree and are likely to comply with the investigator's instructions

Exclusion Criteria:

* Any illness that, in the opinion of the investigator, might confound the results of the study or pose additional risks to the patient
* Use of illicit drugs or over consumption of alcohol (> 3 beers/day)
* Being legally incapacitated, having significant emotional problems at the time of the study

Ages: 12 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Actual)
Dates: Start 2000-06; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
The difference in change in daily insulin need between baseline and month 48, between placebo and ChAgly CD3 treated patients | 48 months

CONTACTS AND LOCATIONS:
Overall Officials: Bart Keymeulen, MD,PhD, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (5):
- Belgium (4):
  - Universitair Ziekenhuis Antwerpen, Antwerp
  - Universitair Ziekenhuis and Diabetes Research Center - Brussels Free University-VUB, Brussels
  - Hopital Erasme, Brussels
  - Department of Endocrinology and Nephrology, UZ Gasthuisberg, Katholieke Universiteit Leuven -KUL, Leuven
- Hopital Schwabbing, Munich, Germany

REFERENCES:
- [Background] Keymeulen B, Vandemeulebroucke E, Ziegler AG, Mathieu C, Kaufman L, Hale G, Gorus F, Goldman M, Walter M, Candon S, Schandene L, Crenier L, De Block C, Seigneurin JM, De Pauw P, Pierard D, Weets I, Rebello P, Bird P, Berrie E, Frewin M, Waldmann H, Bach JF, Pipeleers D, Chatenoud L. Insulin needs after CD3-antibody therapy in new-onset type 1 diabetes. N Engl J Med. 2005 Jun 23;352(25):2598-608. doi: 10.1056/NEJMoa043980. PMID 15972866
- [Derived] Keymeulen B, Walter M, Mathieu C, Kaufman L, Gorus F, Hilbrands R, Vandemeulebroucke E, Van de Velde U, Crenier L, De Block C, Candon S, Waldmann H, Ziegler AG, Chatenoud L, Pipeleers D. Four-year metabolic outcome of a randomised controlled CD3-antibody trial in recent-onset type 1 diabetic patients depends on their age and baseline residual beta cell mass. Diabetologia. 2010 Apr;53(4):614-23. doi: 10.1007/s00125-009-1644-9. Epub 2010 Jan 14. PMID 20225393